CLINICAL TRIAL: NCT05592301
Title: Canadian Patent Foramen Ovale and Perioperative Stroke Evaluation Study (CAPPRES): A Feasibility Study
Brief Title: Patent Foramen Ovale (PFO) and Risk of Perioperative Stroke
Acronym: CAPPRES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Peter Munk Cardiac Centre (Unknown)
Responsible Party: Principal Investigator, Eric Horlick, Director, Structural Heart Disease, University Health Network, Toronto
Other Study IDs: 21-5671; CAPPRES (Other: UHN)
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Patent Foramen Ovale
Keywords: Patent Foramen Ovale; Perioperative Stroke; Diffusion-weighted Magnetic Resonance Imaging
MeSH Terms: conditions — Foramen Ovale, Patent | interventions — Diffusion Magnetic Resonance Imaging; Ultrasonography, Doppler, Transcranial; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical patients: Patients undergoing major non-cardiac, non-vascular, and non-brain surgery who will be examined for a presence of PFO
  Interventions: Diagnostic Test: Diffusion-weighted Magnetic Resonance Imaging (DW-MRI); Diagnostic Test: Transcranial Doppler (TCD); Diagnostic Test: Transthoracic Echocardiogram (TTE)

INTERVENTIONS:
Diagnostic Test: Diffusion-weighted Magnetic Resonance Imaging (DW-MRI) — The Diffusion-weighted Magnetic Resonance Imaging (DW-MRI) is used to diagnose perioperative stroke.
Diagnostic Test: Transcranial Doppler (TCD) — Used to diagnose PFO
Diagnostic Test: Transthoracic Echocardiogram (TTE) — Used to diagnose PFO.

SUMMARY:
This is a multi-centre, prospective cohort study to determine if asymptomatic PFO is a risk factor for developing perioperative overt and covert stroke in patients undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
There is emerging evidence regarding the increased risk of perioperative stroke in patients with PFO, leading to an important clinical practice question: whether PFO should be considered in the perioperative risk assessment in non-cardiac surgery patients. The evidence base, however, comes from retrospective studies with numerous limitations.

Patients referred for general, orthopedic, urological, gynecologic, spinal, or thoracic surgery will be screened and consented during the surgery pre-admission clinic visit, and then undergo PFO screening using transcranial Doppler (TCD) and transthoracic echocardiography (TTE). Patients screened PFO+ (n=102) and matched PFO- controls (n=102) will have DW-MRI between postoperative days 2 and 7. Study personnel will conduct phone surveys at 30-day and 1-year post-surgery to collect data on other clinical outcomes. Patients will also be administered cognitive and patient-reported outcome measures assessments before enrollment, and 30-day and 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. patients 18 years and above;
2. referred for an elective, non-cardiac, non-vascular and non-brain surgery;
3. with an estimated hospital length of stay ≥2 days. We will include patients referred for general, orthopedic, urological, gynecologic, spinal or thoracic surgery.

Exclusion Criteria:

1. patients in need for long-term, perioperative anticoagulants;
2. those with comorbidities that potentially increase the risk of perioperative stroke;
3. contraindications to MRI;
4. unable to complete or adhere to the study.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients referred for an elective, non-cardiac, non-vascular and non-brain surgery
Sampling Method: Non-Probability Sample
Enrollment: 408 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PFO in the target (surgical) population | Pre-operative
  Identifying PFO status using TCD & TTE
The incidence of perioperative stroke in patients without PFO | Within 30 days of surgery
  Identifying perioperative stroke incidence using DW-MRI
Study enrollment rate | Pre-operative
  Establishing study enrollment rate and the reasons for refusals to participate
Proportion of patients completing the DW-MRI test | 2-7 days post surgery
  Developing mechanisms to successfully arrange the DW-MRI within a short timeframe

CONTACTS AND LOCATIONS:
Overall Officials: Eric Horlick, MD, Principal Investigator — University Health Network, Peter Munk Cardiac Centre; Lusine Abrahamyan, MD, PhD, Principal Investigator — University Health Network, Theta Collaborative; Aleksandra Pikula, MD, Principal Investigator — University Heath Network, Division of Neurology
Locations (1):
- Toronto General Hospital, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hobbes B, Akseer S, Pikula A, Huszti E, Devereaux PJ, Horlick E, Abrahamyan L. Risk of Perioperative Stroke in Patients With Patent Foramen Ovale: A Systematic Review and Meta-analysis. Can J Cardiol. 2022 Aug;38(8):1189-1200. doi: 10.1016/j.cjca.2022.02.026. Epub 2022 Mar 3. PMID 35247468